CLINICAL TRIAL: NCT04621071
Title: Evaluation of the Efficacy of Probiotics to Reduce the Duration and Symptoms of COVID-19 (PROVID-19 Study): a Randomized, Double-blind, Controlled Trial
Brief Title: Efficacy of Probiotics in Reducing Duration and Symptoms of COVID-19
Acronym: PROVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-3700
Record Dates: First submitted 2020-11-05; First posted 2020-11-09 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: covid; sars-cov-2; coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Probiotics; stearic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Two probiotic strains will constitute the experimental arm (Probiotics). Patients will take two capsules a day (one closed capsule to swallow and one open capsule mixed with maple syrup) from Day 1 to Day 10 and one closed capsule to swallow from Day 11 to Day 25.They will stop the treatment if they are admitted to the hospital. The treatment will last a maximum of 25 days.
  Interventions: Dietary Supplement: Probiotics (2 strains 10x10^9 UFC)
- Placebo (Placebo Comparator): Potato starch and magnesium stearate will constitute the comparator arm (Placebo). Patients will take two capsules a day (one closed capsule to swallow and one open capsule mixed with maple syrup) from Day 1 to Day 10 and one closed capsule to swallow from Day 11 to Day 25.They will stop the treatment if they are admitted to the hospital. The treatment will last a maximum of 25 days.
  Interventions: Dietary Supplement: Placebo (potato starch and magnesium stearate)

INTERVENTIONS:
Dietary Supplement: Probiotics (2 strains 10x10^9 UFC) — Probiotic vs Placebo (1:1)
  Arms: Probiotics
Dietary Supplement: Placebo (potato starch and magnesium stearate) — Probiotic vs Placebo (1:1)
  Arms: Placebo

SUMMARY:
COVID-19 disease caused by a new coronavirus (SARS-CoV-2) has received worldwide attention. No specific antiviral treatment is recommended for COVID-19 and no vaccine is currently available. Probiotics may be considered as an option of treatment since they have anti-viral effect, trigger immunomodulation and have low side-effects.

This randomized controlled trial aims to evaluate the efficacy of probiotics to reduce the duration and symptoms of COVID-19 in a symptomatic population tested positive to SARS-CoV-2, self-caring at home.

DETAILED DESCRIPTION:
Rational: COVID-19 disease is caused by a new coronavirus (SARS-CoV-2) and has received worldwide attention. No specific antiviral treatment is recommended for COVID-19 and no vaccine is currently available so far. Several strong arguments support the study of probiotics for COVID-19: 1) probiotics act on viruses by various well described mechanisms (reduction of absorption, cellular internalization of the virus, production of metabolites / substances having a direct antiviral effect; and immunomodulation); 2) probiotics are considered with a high level of evidence (meta-analysis) to reduce diarrhea (associated with antibiotics and Clostridium difficile) and for respiratory tract infections; 3) probiotics are affordable and available with low side-effects.

Objectives:

1. Evaluate the effect of probiotics on the duration of COVID-19 in symptomatic patients, with moderate forms of the disease.
2. Evaluate the effect of probiotics on the severity of COVID-19 in symptomatic patients, with moderate forms of the disease.
3. Evaluate the effect of probiotics on the evolution of oral and fecal microbiota in symptomatic patients, with moderate forms of the COVID-19 disease.

Population: Men and women, 18 years or older, with a first positive test for COVID-19 in the last 5 days, having symptoms of the COVID-19, self-caring at home, living in Quebec for the next 60 days, able to take medication alone, with access to a phone or to the Internet.

Material: After providing consent remotely (electronic or recorded by phone), patients will receive by mail at home: : a leaflet explaining the study, the study product (probiotics or placebo) for 25 days, a container of maple syrup and a cup, a thermometer, an oximeter, a logbook, 2 saliva sample self-collection kits, 2 stool sample self-collection kits and instruction sheets.

Randomization: Patients will be randomized in one of the study groups (stratified by age and gender). The randomization is double-blind and uses a ratio 1:1. Group A: will take probiotics for up to 25 days / Group B: will take placebo for up to 25 days.

Follow-up: Upon inclusion in the study, the participant will complete a questionnaire that will focus on socio-demographic (age, marital status), medical (weight, height, general health, current medication, symptoms…), food intake and other relevant information. The participants will fill a daily booklet evaluating their symptoms, compliance to treatment, medication intake, temperature, oxygen saturation value, etc. For those who will be admitted to hospital, data on their admission, complications and treatments will be collected. At 55 days after their enrollment, will fill an end of study questionnaire (symptoms, satisfaction, well-being, etc.).

Samples: The study includes the optional collection of saliva and stool samples twice, on Day 1 (before the first product is taken) and on Day 10.

ELIGIBILITY:
Inclusion Criteria:

* First positive test for COVID-19 in the last 5 days;
* Having symptoms of the COVID-19 at enrollment;
* Self-caring at home;
* Living in Quebec for the next 60 days;
* Able to take medication alone;
* With access to a phone or to the Internet;
* Able to give informed consent.

Exclusion Criteria:

* Taking probiotic supplements at enrollment;
* Taking antibiotics for a reason other than COVID-19 at enrollment;
* Allergies to soy, lactose, yeast, maltodextrin, vitamin C, potato starch, magnesium stearate, hypromellose or titanium dioxide;
* Has a chronically weakened immune system (AIDS, lymphoma, chemo-radio- corticosteroid therapy, immunosuppressive pathology);
* Was treated with chemo-radio-corticosteroid therapy in the last 6 months;
* Has active cancer;
* Taking immunosuppressive drugs (e.g. anti-rejection treatment after organ transplant);
* Already participating in another clinical trial;
* Is pregnant, expects to become pregnant in the next few months or is breastfeeding;
* Has any other condition that would prevent safe participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Duration of symptoms of the COVID-19 | During the period of the treatment (from Day 1 to Day 25)
  Number of days before symptoms disappear

SECONDARY OUTCOMES:
Severity of the COVID-19 | During the period of the study, first day in (at randomization) to last day in (last follow-up 30 days after the end of treatment) (from Day 1 to Day 55)
  Categorical distribution among: 1) at home without symptoms, 2) at home with symptoms, 3) hospitalized without O2 supplementation, 4) hospitalized with O2 supplementation, 5) admitted to intensive care unit, 6) deceased
Evolution of oral and fecal microbiota | At Day 1 (baseline) and Day 10 of the treatment
  Metagenomic sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Pasquier, Dr, Principal Investigator — CIUSSSE-CHUS
Locations (1):
- CIUSSS de L'Estrie-CHUS Hospital, Sherbrooke, Quebec, Canada